CLINICAL TRIAL: NCT02050503
Title: Ability of Intranasal Transmucosal Fentanyl Pectin Nasal Spray to Prevent Breakthrough Pain Episodes in Patients With Radiation-induced Oropharyngeal Mucositis
Brief Title: Intranasal Transmucosal Fentanyl Pectin for Breakthrough Cancer Pain in Radiation-induced Oropharyngeal Mucositis
Acronym: CP073
Status: Completed | Type: Observational
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Sponsor
Other Study IDs: CP073
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Breakthrough Pain; Mucositis; Radiotherapy; Chemotherapy; Head and Neck Cancer
Keywords: Mucositis; Breakthrough pain; Head Nad neck cancer; Intranasal transmucosal fentanyl in pectin
MeSH Terms: conditions — Breakthrough Pain; Mucositis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- intranasal transmucosal fentanyl pectin: intranasal transmucosal fentanyl in pectin (100, 200, 400 or 800 microg) intranasal route titration phase 7 days treatment phase until completing treatment of 12 consecutive episodes of breakthrough pain

SUMMARY:
An open-label, non-randomized study to assess the titration, safety and efficacy of intranasal fentanyl pectin nasal spray for the treatment of secondary breakthrough pain secondary to radiation-induced mucositis in patients with confirmed tolerance of opioid therapy for chronic pain.

Study objectives include assessment of breakthrough pain episodes related with food intake in patients with mucositis secondary to radiotherapy or radio-chemotherapy for head and neck tumors

DETAILED DESCRIPTION:
An open, non-randomized study design was used to assess the titration, safety and efficacy of intranasal fentanyl in pectin for the treatment of secondary breakthrough pain in patients with confirmed tolerance of opioid therapy for chronic pain secondary to radiation-induced mucositis. The study plans to include 30 evaluable patients from multiple centers throughout the country. The trial comprises a screening period, an open titration period, and an open-label treatment period in which at least 12 breakthrough pain episodes are to be treated.

ELIGIBILITY:
Inclusion Criteria:

A histologically confirmed diagnosis of head and neck carcinoma Treatment in the form of radiotherapy or radio-chemotherapy Breakthrough pain related to swallowing (one to four daily episodes) Treatment with controlled release opioids at the time of inclusion: at least 60 mg of morphine sulfate daily, at least 25 microg of transdermal fentanyl per hour, at least 30 mg of oral oxycodone daily, at least 8 mg of oral hydromorphone daily

Exclusion Criteria:

* Patients without controlled release opioid treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults of either sex and over 18 and under 75 years of age, receiving continued treatment with long half-life or controlled release opioids, experiencing breakthrough pain secondary to mucositis in the context of radiotherapy or radio-chemotherapy for head and neck tumors.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Difference | 30 minutes after PecFent administration
  Pain Intensity difference: Pain Intensity will be measured 30 min after starting food intake during the screening phase and 30 min after intranasal transmucosal fentanyl in pectin administration/food intake during the treatment phase

SECONDARY OUTCOMES:
number of episodes of breakthrough pain requiring additional (rescue) analgesic treatment after administration of the study medication | 12 episodes of breakthrough pain presenting within a maximum of 7 days.
  The number of episodes of breakthrough pain requiring additional (rescue) analgesic treatment after administration of the study medication.
  Patient rating of drug efficacy measured on a scale from 0 to 10 (0 = ineffective, 10 = totally effective).
  Quality of life assessed with the European Organization for Research and Treatment of Cancer quality of life questionnaire -INF025 in its validated Spanish version, administered on the screening visit and at the end of the study.
  Patient rating of drug ease of use measured on a scale from 1 to 4 (1 = very complicated, 4 = very simple).

OTHER OUTCOMES:
safety of intranasal transmucosal fentanyl | 7 days
  The appearance of adverse effects during the study Physical examination at each visit Vital signs: blood pressure, pulse Concomitant medication for breakthrough pain Reasons for patient study withdrawal (in the event of withdrawal)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro De la Torre, MD, Principal Investigator — GICOR & Hospital Puerta de Hierro
Locations (1):
- Alejandro de la Torre. Hospital Puerta de Hierro, Majadahonda, Madrid, Spain